CLINICAL TRIAL: NCT05267444
Title: The Effects of a Tele-health Program to Facilitate the Usage of Internet of Things Among Community-dwelling Frail Older Adults: a Randomized Controlled Trial
Brief Title: The Effects of a Tele-health Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0036805
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Frailty; Old Age; Debility
Keywords: technology device; occupational therapy; young adult; frail older adults; self-care
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Individualized motion-based interactive game program
  Interventions: Procedure: Individualized motion-based interactive game program
- Control group (No Intervention): The control group participants will receive usual care, that is, service that provided by community elderly center

INTERVENTIONS:
Procedure: Individualized motion-based interactive game program — The participants will receive a 12-session, 4.5 months home visit service that is provided by the young adults, and supervised by an occupational therapist. Young adults will follow the individualized exercise plan with the older adults, facilitate their use of interactive games, provide psychological and technological support to help older adults cope with their fear of using technologies to perform physical activity.
  Arms: Intervention group

SUMMARY:
Frailty is a state of being vulnerable and functional disable due to age-related decline of multiple physiological systems, and is often associated with higher risk of falls, institutionalization, hospitalization, disability, dementia, and death. One of the best strategies to combat the burden of frailty is to promote physical activity in the aging population, especially to the older adults who are already in a frail condition

ELIGIBILITY:
For older adults:

Inclusion Criteria:

* aged 60 or above
* having level of frailty from "managing well" to "living with severe frailty" (Clinical Frailty Scale score 3-7) -- HK-MoCA score 23 or less (add one point to people who had less than 6 year formal education and add 2 points to people who had no formal education)

Exclusion Criteria:

* currently receiving any kind of rehabilitation service
* living with another older adult who is participating in the same study.

For young adults:

Inclusion Criteria:

* aged 17 to 35
* having educational level of secondary 5 or above

Exclusion Criteria:

- having a full-time job

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
The change of physical activity before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Physical activities of the older adults will be measured by the Chinese version of the Physical Activity Scale for the Elderly. The PASE-C is a 12-items scale estimating the frequency and intensity of older adults' lifestyle physical activities with three types of physical activities (leisure-time activity: 5 items; household activity: 6 items; work-related activity: 1 item) during the previous 7-day period. The total score is computed by the multiplication on the time spent (recorded as never, seldom: 1-2 days per week, sometimes: 3-4 days per week, and often: 5-7 days per week) or participation (yes/no) on each activity by items weights, and summarize all the items. Higher scores mean higher frequency and intensity of physical activities.

SECONDARY OUTCOMES:
The change of balance before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Balance will be assessed using the Berg functional balance scale. It is a 14-item scale designed to measure balance of the older adult in a community setting. The scores of the scale range from 0 to 56, with higher the score, better the balance
The change of cognition status before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Cognition status will be measured by the Chinese version of the Mini-Mental State Examination. The Mini mental state examination contains questions in seven domains, such as temporal and spatial orientation, word encoding, attention and calculation, word recall, language, and visual constructive capacity. The scores of scale range from 0 to 30, with higher scores indicate better cognitive status
The change of short-term memory before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Short-term memory will be assessed using the digit span forward test. It consists of the presentation of a list of numbers, which should be correctly repeated in a forward order immediately after their presentation. Higher scores mean better short-term memory.
The change of loneliness level before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Loneliness will be assessed using the UCLA Loneliness Scale. Each participant will be asked the following three questions: "How often do you feel that you lack companionship?", "How often do you feel left out?" and "How often do you feel isolated from others?". Each question had three options to reflect the frequency:1 = Hardly ever, 2 = Some of the time, and 3 = Often). The values for each question will be summed to get a loneliness score ranging from 3 to 9, with higher values indicating greater loneliness.
The change of social isolation before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Social isolation will be measured by the two subscales of the 6-item Lubben Social Network Scale-6. Each subscale score ranges from 0 to 15, with lower score indicating greater isolation.
The change of quality of life before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Quality of life will be measured by SF-12v2, which has been translated, validated and proven reliable for use among the Hong Kong Chinese population. Score 50 is a norm globally. Higher score means better quality of life.
The change of depression level before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Depression will be measured by the Chinese version of the Geriatric Depression Scale. The scale ranges from 0-12, with higher score indicates higher depression level.
The change of self-efficacy before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Self-efficacy will be assessed using the Chinese version of the General Self-Efficacy Scale. It is a ten-item scale measuring a broad and stable sense of personal competence to deal efficiently with a variety of stressful situations. The C-GSE measures the strength dimension of self-efficacy on a four-point Likert scale. Scores are summed to give a total range from 10 to 40; higher scores represent greater self-efficacy.
The change of social connectedness before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Social connectedness will be assessed using the Social Connectedness Scale-Revised. The SCS-R, like its predecessor, measures social connectedness as a psychological sense of belonging or, more specifically, as a cognition of enduring interpersonal closeness with the social world in toto. The scale consists of 20 items (10 positive and 10 negative) rated on a 6-point Likert scale with higher scores represent better social connectedness
The change of attitude towards elderly before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Attitude towards elderly will be assessed using Kogan's (1961) Attitude toward Old People scale. The Attitude toward old people scale consists of 34 items grouped into two factors that assess positive and negative attitudes toward old people. Kogan's attitude toward old people consisted of 3 domains: personal appearance, resemblance, and the nature of interpersonal relations across age generations. The scores of the scale range from 34 to 204, with higher scores mean better attitude towards elderly
The change of life satisfaction before and after the program | baseline pre-intervention, 4.5 months when the program is completed
  Life satisfaction will be assessed using the satisfaction with life scale (SWLS).It is a 5-item scale designed to measure global cognitive judgments of one's life satisfaction (not a measure of either positive or negative affect). Participants will indicate how much they agree or disagree with each of the 5 items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. Higher scores indicate better life satisfaction
The change of community involvement before and after the completion of the program | Six months after the completion of the program
  Community involvement will be assessed by asking the participants their number of hours involved in elderly services six months after the completion of the program. Higher hours represent better community involvement
Recruitment rate after the completion of the program | 6 months after the completion of the program
  Recruitment rate will be obtained by asking the participant their working status at 6 months after the completion of the program. More people recruited to elderly service work, better the recruitment rate

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, Ph.D., Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Community center, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No